CLINICAL TRIAL: NCT00055146
Title: A Multicenter, Phase II Study of ONTAK (Denileukin Diftitox) in Patients With Previously-Treated Chronic Lymphocytic Leukemia
Brief Title: Study of ONTAK in Patients With B-Cell Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L4389-34
Record Dates: First submitted 2003-02-19; First posted 2003-02-21 (Estimated); Last update posted 2009-04-17 (Estimated); Status verified 2009-04

CONDITIONS: Leukemia, Lymphocytic, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — denileukin diftitox

INTERVENTIONS:
Drug: ONTAK

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of ONTAK in previously treated patients with chronic lymphocytic leukemia (CLL)

ELIGIBILITY:
Inclusion Criteria:

* Patients with B-cell Chronic Lymphocytic Leukemia, Rai Stage 0-II with indication for treatment by NCI Working Group Criteria or Rai Stage III or IV.
* Patients must have received at least one prior purine analogue-based chemotherapy regimen.
* ECOG Performance Status of 0, 1, or 2.
* Female patients cannot be pregnant and must use birth control during the course of the study and for three weeks after the study ends.

Exclusion Criteria:

* Prior treatment with ONTAK (DAB389IL-2) or DAB486IL-2.
* Received any therapy for CLL within 35 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2003-03; Primary Completion 2006-03 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Objective Clinical Response

SECONDARY OUTCOMES:
Time-to-Progression
Duration of response

CONTACTS AND LOCATIONS:
Overall Officials: Elyane Lombardy, M.D., Study Director — Ligand Pharmaceuticals
Locations (14):
- United States (5):
  - Pacific Coast Hematology/Oncology Medical Group, Inc., Fountain Valley, California
  - UCSD School of Medicine, La Jolla, California
  - Rush-Presbyterian St. Luke's Cancer Center, Chicago, Illinois
  - Weill Medical College of Cornell University/New York Presbyterian Hospital, New York, New York
  - University of Texas, M.D. Anderson Cancer Center, Houston, Texas
- Montecaseros, Mendoza, Argentina
- Australia (2):
  - Peter MacCallum Cancer Institute, East Melbourne, Victoria
  - Oncology Day Unit, Frankston Hospital, Frankston
- Brazil (5):
  - Hospital Araujo Jorge - Associacao de Combate ao Cancer em Goias, Goiânia, Goiás
  - Hospital de Clinicas da Universidade Federal do Parana, Curitiba, Paraná
  - Universidade Federal do Rio de Janeiro - Hospital Universitario Clementino Fraga Filho, Rio de Janeiro, Rio de Janeiro
  - Hospital de Cancer de Barretos - Fundacao Pio XII, Barretos, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo
- Sir Mortimer B. Davis - Jewish General Hospital, Montreal, Quebec, Canada